CLINICAL TRIAL: NCT03656783
Title: Effects of Biectegravir-Emtricitabine-Tenofovir Alafenamide on Coronary Flow Reserve in Stable HIV Patients (B/F/TAF-CFR) - Pilot Study
Brief Title: Effects of Biktarvy on CFR in Stable HIV Patients
Acronym: BETTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Tufts Medical Center (Other); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Marcelo F. Di Carli, MD, FACC, Chief of Nuclear Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001579
Record Dates: First submitted 2018-08-31; First posted 2018-09-04 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: HIV
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; bictegravir; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HIV patients on stable therapy (Other): HIV patients on stable therapy switching from Abacavir/Lamivudine/Dolutegravir (ABC/3TC/DTG) to the Bictegravir/ Emtricitabine/Tenofovir Alafenamide (B/F/TAF)
  Interventions: Drug: Biktarvy

INTERVENTIONS:
Drug: Biktarvy — Open-label, multicenter, single-arm study to Evaluate the Safety and Efficacy of Switching from Regimens Consisting of Abacavir/Lamivudine/Dolutegravir (ABC/3TC/DTG) to the Bictegravir/ Emtricitabine/Tenofovir Alafenamide (B/F/TAF) Fixed-Dose Combination (FDC) in Virologically-Suppressed HIV-Infected Adult Subjects
  Other Names: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF)

SUMMARY:
Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) is a single pill regimen that was approved by the FDA in February 2018 for treatment of HIV. The marketed name of the drug is Biktarvy. In two phase 3 comparative clinical trials, including one with ABC/3TC/DTG, it was found to be non-inferior to dolutegravir-containing regimens in terms of virologic outcomes. B/F/TAF was also well tolerated, with few discontinuations for adverse events. As a result, B/F/TAF is an ideal non-abacavir containing regimen to assess the effect of removing ABC on coronary flow reserve.

DETAILED DESCRIPTION:
Positron emission tomography (PET) imaging allows precise and reproducible quantification of myocardial blood flow, thereby providing a direct assessment of coronary vascular health. Coronary flow reserve (CFR, calculated as the ratio of peak hyperemic myocardial blood flow over that at rest) is emerging as a powerful quantitative prognostic imaging marker of clinical cardiovascular risk. CFR provides a robust and reproducible clinical measure of the integrated hemodynamic effects of epicardial coronary artery disease (CAD), diffuse atherosclerosis, vessel remodeling, and microvascular dysfunction resulting from endothelial cell dysfunction on myocardial tissue perfusion across the entire coronary circulation. These processes have direct relevance to the underlying vascular pathobiology in patients with HIV infection. Consequently, quantitative CFR provides a unique opportunity to examine the potential impact of novel therapies on the biology of the disease and its association with cardiovascular outcomes. By testing the fundamental concept of whether novel ART therapies in HIV can lead to improved coronary blood flow and myocardial tissue perfusion, TAF-CFR would provide important mechanistic insights of the capabilities of TAF therapy to improve key determinants of clinical risk.

This is an open label, multicenter, uncontrolled, single arm pilot study. Patients with stable HIV currently treated with abacavir/lamivudine/dolutegravir STR regimens will be eligible for the B/F/TAF-CFR study. PET scans will be performed after enrollment while on the abacavir/lamivudine/dolutegravir STR regimen and at 24 weeks after the switch to B/F/TAF regimen. Patients will be encouraged to remain on stable medical therapy throughout the enrollment period.

ELIGIBILITY:
Inclusion Criteria:

Patients with HIV on abacavir/lamivudine/dolutegravir STR regimens for at least 1 year fulfilling the following inclusion criteria:

1. age ≥ 45 years for men and ≥ 55 years for women;
2. at least one coronary risk factor including smoking, dyslipidemia, hypertension, obesity (BMI >30) or diabetes, or a calculated 10-year risk of heart attack of 7.5% or higher;
3. HIV RNA < 200 copies/mL at last clinical measurement, done within the past 12 months prior to screening, with no intervening HIV RNA > 200;
4. Screening HIV RNA < 50 copies/mL, CBC, and chemistries that, in the judgment of the investigator, do not preclude the use of Biktarvy.

Exclusion Criteria:

1. patients not fulfilling inclusion criteria;
2. unstable HIV disease or other medical condition that, in the opinion of the investigator, would interfere with the conduct of the study;
3. history of cardiomyopathy (LVEF <40%) or significant valvular heart disease;
4. cirrhosis;
5. end stage renal disease on dialysis;
6. uncontrolled hypertension (defined as SBP >200 or DBP >110);
7. pregnancy;
8. Patients requiring medications contraindicated with the components of B/F/TAF;
9. Patients on active treatment for severe asthma or severe COPD.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Di Carli, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huck DM, Weber B, Parks S, Divakaran S, Brown JM, Bibbo CF, Barrett L, Hainer J, Bay C, Martell L, Kogelman L, Triant VA, Chu J, Lin NH, Melbourne K, Sax PE, Di Carli MF. Coronary Microcirculatory Dysfunction in People With HIV and Its Association With Antiretroviral Therapy. J Am Heart Assoc. 2023 Nov 21;12(22):e029541. doi: 10.1161/JAHA.123.029541. Epub 2023 Nov 10. PMID 37947105

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV Patients on Stable Therapy: Patients with stable HIV treated with abacavir/lamivudine/dolutegravir STR regimens switching to B/F/TAF-CFR
Period: Overall Study
Arm/Group | HIV Patients on Stable Therapy
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HIV Patients on Stable Therapy
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.44 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Global CFR
Description: Change in global coronary flow reserve, as measured by PET imaging at baseline and 24 weeks after initiation of B/F/TAF therapy.
  Coronary flow reserve (CFR), the ratio of peak vasodilator stress to rest myocardial blood flow (MBF), represents the maximal ability to augment coronary flow and myocardial perfusion. Absolute MBF was computed from the rest and stress myocardial perfusion PET images using commercially available software (Corridor4DM; Ann Arbor, Michigan) and a two-compartment tracer kinetic model. Impaired MBFR is defined as a ratio of <2.0, which is associated with increased cardiovascular risk.
Time Frame: baseline and week 24
Population: We enrolled men 45 years and over and women 55 years and over with HIV who were stable on a DTG/3TC/ABC regimen with virologic suppression for at least one year, and with at least one coronary risk factor (current smoking, dyslipidemia, hypertension, diabetes, obesity, or a calculated 10-year predicted risk of cardiovascular events of 7.5 percent or over) but without overt cardiovascular disease.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | HIV Patients on Stable Therapy
Number analyzed (Participants) | 25
ratio | -.05 [-.25 to 0.15]

2. Secondary Outcome: Change in Peak Stress Global MBF
Description: Change (from baseline) in peak-stress global myocardial blood flow (in mL/min/g) at 24 weeks after initiation of B/F/TAF.
  Absolute MBF was computed from the rest and stress myocardial perfusion PET images using commercially available software (Corridor4DM; Ann Arbor, Michigan) and a two-compartment tracer kinetic model. Impaired stress MBF is defined as <1.8 mL/min/g and is associated with increased cardiovascular risk.
Time Frame: baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: mL/min/g
Arm/Group | HIV Patients on Stable Therapy
Number analyzed (Participants) | 25
mL/min/g | 0.09 [-.05 to .23]

3. Secondary Outcome: Change in Serum Biomarkers of Inflammation (Hs-CRP (in mg/L))
Description: Change in serum biomarkers of inflammation (hs-CRP (in mg/L)) at 24 weeks after initiation of B/F/TAF.
  Serum biomarkers of inflammation (high sensitivity C-reactive protein) were measured. hs-CRP > 1 mg/L are considered abnormal and associated with increased cardiovascular risk.
Time Frame: Baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | HIV Patients on Stable Therapy
Number analyzed (Participants) | 25
mg/L | -0.40 [-1.52 to 0.72]

4. Secondary Outcome: Change in Myocyte Injury and Strain (hs Troponin (in ng/L))
Description: Change in Myocyte Injury and Strain (hs Troponin (in ng/L)) at 24 weeks after initiation of B/F/TAF.
  Serum biomarkers of myocardial injury/strain (high sensitivity troponin) were measured. hs-troponin >14 ng/L are considered abnormal and associated with increased cardiovascular risk.
Time Frame: Baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: ng/L
Arm/Group | HIV Patients on Stable Therapy
Number analyzed (Participants) | 25
ng/L | -0.04 [-1.11 to 1.02]

5. Secondary Outcome: Change in Myocyte Injury and Strain (NT-proBNP (in pg/mL))
Description: Change in Myocyte Injury and Strain (NT-proBNP (in pg/mL)) at 24 weeks after initiation of B/F/TAF.
  Serum biomarkers of myocardial injury/strain (NT-pro-BNP) were measured. NT-proBNP > 100 pg/mL are considered abnormal and associated with increased cardiovascular risk.
Time Frame: Baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | HIV Patients on Stable Therapy
Number analyzed (Participants) | 25
pg/mL | -14.2 [-43.4 to 15.2]

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from consent through 24-week End of Treatment visit.
Groups:
- HIV Patients on Stable: HIV patients on stable therapy switching from Abacavir/Lamivudine/Dolutegravir (ABC/3TC/DTG) to the Bictegravir/ Emtricitabine/Tenofovir Alafenamide (B/F/TAF)
Arm/Group | HIV Patients on Stable
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Patients on Stable (N=25)
Shortness of Breath (Cardiac disorders) | 2 (2) — Subjects experienced shortness of breath in response to Regadenoson stress test.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03656783/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT03656783/ICF_001.pdf